CLINICAL TRIAL: NCT01230086
Title: hs Troponin Release in Relation to Different ICD-Implantation Procedures
Brief Title: Trop-Shock DFT-testing Versus None
Acronym: Trop-Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-005
Record Dates: First submitted 2010-10-26; First posted 2010-10-28 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Defibrillation Testing - ICD Therapy Optimisation
Keywords: ICD; DFT-testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICD implantation only (Active Comparator): ICD Implantation without testing of defibrillation threshold testing
  Interventions: Device: ICD Implantation without DFT testing; Device: T-wave shock with induction of ventricular fibrillation
- Modified upper limit of vulnerability testing (Active Comparator): Modified testing of "upper limit of vulnerability"
  Interventions: Device: Upper limit of vulnerability testing
- VF-Induction (Active Comparator): traditional VF-induction with T-Wave shock
  Interventions: Device: T-wave shock with induction of ventricular fibrillation

INTERVENTIONS:
Device: ICD Implantation without DFT testing — Implantation
  Arms: ICD implantation only
Device: Upper limit of vulnerability testing — Upper limit of vulnerability testing
  Arms: Modified upper limit of vulnerability testing
Device: T-wave shock with induction of ventricular fibrillation — Traditional safety margin testing for defibrillation threshold
  Arms: ICD implantation only; VF-Induction

SUMMARY:
Implantation of a cardioverter defibrillator (ICD) is the treatment of choice for primary and secondary prevention of sudden cardiac death. Traditionally, intraoperative testing for sensing and defibrillation capabilities of the ICD system is performed. Modern implantation strategies suggest a non-testing approach because net-benefit of a testing versus a non-testing strategy is questionable and because arrhythmia induction and defibrillation may cause micro damage to the heart.

The study aims to investigate the contribution of different steps in the ICD implantation procedure (implantation of the lead, shock delivery and induced ventricular fibrillation) with respect to their potential damage to the heart measured by high sensitivity (HS) TroponinT.

ELIGIBILITY:
Inclusion Criteria:

* ICD-Implantation in patients with coronary artery disease or dilative cardiomyopathy

Exclusion Criteria:

* Atrial fibrillation with inappropriate anticoagulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-08; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Influence of different ICD-implantation strategies on release of high sensitivity Troponin | 6 hours

SECONDARY OUTCOMES:
Influence of different ICD-implantation strategies on BNP release | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität München, München, Bavaria, Germany

REFERENCES:
- [Derived] Semmler V, Biermann J, Haller B, Jilek C, Sarafoff N, Lennerz C, Vrazic H, Zrenner B, Asbach S, Kolb C. ICD Shock, Not Ventricular Fibrillation, Causes Elevation of High Sensitive Troponin T after Defibrillation Threshold Testing--The Prospective, Randomized, Multicentre TropShock-Trial. PLoS One. 2015 Jul 24;10(7):e0131570. doi: 10.1371/journal.pone.0131570. eCollection 2015. PMID 26208329
- See also: Publication Trop-Shock-Study — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0131570